CLINICAL TRIAL: NCT05034120
Title: A Study to Investigate the Food Effect on the Pharmacokinetics of XZP-3621 Tablets and the Absorption, Metabolism and Excretion of XZP-3621 in Chinese Healthy Volunteers
Brief Title: Food Effect and Mass Balance Study of XZP-3621 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XZP-3621-1002
Record Dates: First submitted 2021-08-19; First posted 2021-09-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: XZP-3621; Food-Effect; Mass Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- MB:Single arm (Experimental): 10 subjects will be enrolled in this arm. The subjects will take a single dose XZP-3621 tablet after a low-fat meal and perform excretion collection consistently.
  Interventions: Drug: XZP-3621
- FE:Arm A (Experimental): Cycle1 Day1: fasting; Cycle2 Day10: High-fat meal; Cycle3 Day19: Low-fat meal
  Interventions: Drug: XZP-3621
- FE:Arm B (Experimental): Cycle1 Day1: High-fat meal; Cycle2 Day10: Low-fat meal; Cycle3 Day19: fasting
  Interventions: Drug: XZP-3621
- FE:Arm C (Experimental): Cycle1 Day1: Low-fat meal; Cycle2 Day10: fasting; Cycle3 Day19: High-fat meal
  Interventions: Drug: XZP-3621
- FE:Arm D (Experimental): Cycle1 Day1: fasting; Cycle2 Day10: Low-fat meal; Cycle3 Day19: High-fat meal
  Interventions: Drug: XZP-3621
- FE:Arm E (Experimental): Cycle1 Day1: High-fat meal; Cycle2 Day10: fasting; Cycle3 Day19: Low-fat meal
  Interventions: Drug: XZP-3621
- FE:Arm F (Experimental): Cycle1 Day1: Low-fat meal; Cycle2 Day10: High-fat meal; Cycle3 Day19:fasting
  Interventions: Drug: XZP-3621

INTERVENTIONS:
Drug: XZP-3621 — Administer a single dose of XZP-3621 tablet after a low-fat meal.
  Arms: MB:Single arm
Drug: XZP-3621 — Cycle1(D1-D9): Administer the XZP-3621 tablet on an empty stomach in a single dose on Day1; Cycle2(D10-D18): Administer the XZP-3621 tablet after a high-fat meal in a single dose on Day10; Cycle3(D19-D27): Administer the XZP-3621 tablet after a standard meal in a single dose on Day19.
  Arms: FE:Arm A
Drug: XZP-3621 — Cycle1(D1-D9) : Administer the XZP-3621 tablet after a high-fat meal in a single dose on Day1; Cycle2(D10-D18): Administer the XZP-3621 tablet after a standard meal in a single dose on Day10; Cycle3(D19-D27): Administer the XZP-3621 tablet after on an empty stomach in a single dose on Day19.
  Arms: FE:Arm B
Drug: XZP-3621 — Cycle1(D1-D9): Administer the XZP-3621 tablet after a standard meal in a single dose on Day1; Cycle2(D10-D18): Administer the XZP-3621 tablet on an empty stomach in a single dose on Day10; Cycle3(D19-D27): Administer the XZP-3621 tablet after a high-fat meal in a single dose on Day19.
  Arms: FE:Arm C
Drug: XZP-3621 — Cycle1(D1-D9) : Administer the XZP-3621 tablet on an empty stomach in a single dose on Day1; Cycle2(D10-D18): Administer the XZP-3621 tablet after a standard meal in a single dose on Day10; Cycle3(D19-D27): Administer the XZP-3621 tablet after a high-fat meal in a single dose on Day19.
  Arms: FE:Arm D
Drug: XZP-3621 — Cycle1(D1-D9): Administer the XZP-3621 tablet after a high-fat meal in a single dose on Day1; Cycle2(D10-D18): Administer the XZP-3621 tablet on an empty stomach in a single dose on Day10; Cycle3(D19-D27): Administer the XZP-3621 tablet after a standard meal in a single dose on Day19.
  Arms: FE:Arm E
Drug: XZP-3621 — Cycle1(D1-D9): Administer the XZP-3621 tablet after a standard meal in a single dose on Day1; Cycle2(D10-D18): Administer the XZP-3621 tablet after a high-fat meal in a single dose on Day10; Cycle3(D19-D27): Administer the XZP-3621 tablet on an empty stomach in a single dose on Day19.
  Arms: FE:Arm F

SUMMARY:
This is a single-center, open-label, single-dose phase I study, the study is divided into two stages. The stage 1 is to investigate the absorption, metabolism and excretion of XZP-3621 tablets in healthy Chinese subjects. The stage 2 is to evaluate the effect of food on the Pharmacokinetics of single-dose XZP-3621 tablets in Chinese Healthy Volunteers. In addition, the safety of XZP-3621 tablets in Chinese Healthy Volunteers will also be evaluated.

DETAILED DESCRIPTION:
Stage 1: 10 healthy adult subjects will be included in the study. Excretion (feces, urine) and vomit samples will be collected daily and tested for prototype drug and metabolites of XZP-3621, the metabolites will be identified in all substrates except vomits pose-dose of 400 mg XZP-3621 tablets.

Vomit samples collection: Time interval for subject vomit collection (if any) (planned):0~4 h,4~8 h,8~12 h,12~24 h,24~48 h,48~72 h,72~96 h,96~120 h,120~144 h,144~168 h,168~192 h after taking single XZP-3621 tablet. Samples of all vomits during that time interval will be collected at each time interval after taking single XZP-3621 tablet.

Urine samples collection: Time interval for sample collection(planned):24h before taking single XZP-3621 tablet,0~4 h,4~8 h,8~12 h,12~24 h,24~48 h,48~72 h,72~96 h,96~120 h,120~144 h,144~168 h,168~192 h after taking single XZP-3621 tablet, Urine samples were collected from each subject at a total of 12 time intervals (Only one urine sample should be collected within 24 hours before taking single XZP-3621 tablet), Urine volume was accurately recorded for each time period.

Feces samples collection: Interval of fecal sample collection of subjects (planned):24h before taking single XZP-3621 tablet,0~24 h,24~48 h,48~72 h,72~96 h,96~120 h,120~144 h,144~168 h,168~192 h after taking single XZP-3621 tablet. Feces samples will be collected from each subject at a total of 9 time intervals (Only one sample was collected within 24 h before taking single XZP-3621 tablet), And accurate fecal weight will be recorded for each time period.

PK blood sample collection: PK blood samples of subjects will be collected before administration (within 2 h before administration) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 192 h after administration at 18 collection points. Plasma samples for metabolite identification should be separately packaged.

Stage 2: This stage of study will be a randomized, open, three-cycle crossover study to evaluate the pharmacokinetic effects and safety of a single oral dose of XZP-3621 in healthy subjects on a high-fat diet versus a standard diet.

In this study stage, 24 healthy subjects meeting the requirements of the protocol will be planned to be enrolled and randomly divided into groups A, B, C, D, E and F at 1:1:1:1:1:1 , with 4 subjects in each group. Each subject will undergo three cycles of fasting administration, high-fat postprandial administration, and standard postprandial administration (in random order) throughout the study.

PK blood sample collection: PK blood samples will be collected before taking single XZP-3621 tablet (within 2 h before drug administration) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 192 h after taking single XZP-3621 tablet in each cycle, with a total of 18 collection points.

ELIGIBILITY:
Inclusion Criteria:

* Subject who meet all of the requirements as follows will be included.

  1. Healthy male or female subjects aged 18 to 65 (including 18 and 65);
  2. Male weight ≥50 kg, female weight ≥45 kg, body mass index in the range of 18-28 kg/m2 (including 18 and 28);
  3. No medical history of mental abnormalities, cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system or metabolic abnormalities;
  4. Subjects agree to use effective contraceptive methods, such as condoms, contraceptive sponges, contraceptive gels, contraceptive membrane, intrauterine device, oral or injectable contraceptives, subcutaneous implants, or other contraceptive methods, from screening (2 weeks prior to screening for female subjects) to 6 months after the last dose;
  5. The subject can have a good communication with the investigators, understand and comply with the requirements of this study, understand and sign the informed consent voluntarily.

Exclusion Criteria:

* Subject who meet either of the requirements as follows will be excluded.

  1. Hypersensitivity (hypersensitivity to two or more substances) or known hypersensitivity to XZP-3621 tablets/similar drugs;
  2. Abnormal examination during the screening period with clinical significance (to be determined by the investigator);
  3. Frequent use of sedatives、sleeping pills or other addictive drugs et al;
  4. Those who had a history of drug abuse or urine drug abuse screening positive within 12 months before enrollment;
  5. Smoking more than 5 cigarettes a day, or failing to stop using any tobacco products during the test period;
  6. Positive breath test for alcohol or regular drinkers in the 6 months prior to entry, i.e. drinking more than 3 units per day or more than 21 units per week (one unit is equivalent to a 350 mL bottle of beer or 120 mL of liquor or 30 mL of spirits (over 50°));
  7. Take any prescription medicine or Chinese herbal medicine within 4 weeks before enrollment, and/or Take any over-the-counter (OTC) drug or food supplement (including vitamins, calcium tablets and other health care products) within 2 weeks before the first administration of XZP-3621 tablet;
  8. Those who have participated in other clinical trials and taken experimental drugs within 3 months before enrollment;
  9. Blood donation (including component blood donation) or blood loss of 400 mL within 3 months before enrollment, or blood transfusion;Blood donation (including component blood donation) or blood loss of 200 mL within 1 month before the test;
  10. Have a history of major disease or major surgery or trauma 3 months before screening;
  11. A history of gastrointestinal disease causing clinically significant symptoms such as nausea, vomiting, diarrhea, or malabsorption syndrome, or a history of severe vomiting or diarrhea within the week prior to enrollment;
  12. Female subjects during pregnancy and lactation and female subjects of childbearing age who cannot use contraception as required;
  13. Hepatitis B surface antigen positive, hepatitis C antibody positive, syphilis antibody positive, HIV antibody positive;
  14. Have special dietary requirements (including lactose intolerance) and fail to comply with the provided diet and corresponding regulations;
  15. Subjects who are Dysphagia;
  16. Subjects who refuse to stop any beverage or food containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, grapefruit and beverages containing this ingredient, etc.) 48 hours prior to first administration of XZP-3621 tablets until the end of the study.
  17. Subjects who will refuse to discontinue any CYP3A4 inhibitors and inducers judged by the investigator within 7 days prior to the first administration of XZP-3621 tablets or within 5 half-lives of CYP3A4 inhibitors and inducers (whichever is longer) until the end of the study;
  18. Subjects who are Inability to tolerate venipuncture or poor vascular status;
  19. Subjects who are unsuitable to participate in this study judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
AUC0-t(area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 192 hours
  Pharmacokinetic Data Analysis for XZP-3621 and its metabolites
Cmax(maximum measured concentration of the analyte in plasma) | up to 192 hours
  Pharmacokinetic Data Analysis for XZP-3621 and its metabolites
AUC0-∞(area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 192 hours
  Pharmacokinetic Data Analysis for XZP-3621 and its metabolites
to determine the Mass Balance recovery of orally administered XZP-3621 and its metabolites in all (urine, faeces and vomits) amount excreted (Ae) expressed as a percentage of the administered dose (%Ae) | MB stage:Day1-Day9
  cumulative excretions after a single dose of XZP-3621 and its metabolites in urine, feces and vomits.

SECONDARY OUTCOMES:
Tmax(the time from dosing at which Cmax was apparent) | up to 192 hours
  Pharmacokinetic Data Analysis for XZP-3621 and its metabolites
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | MB Stage:28±3 days,FE Stage:47±3 days
  Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE 5.0
T1/2(Apparent terminal elimination half-life ) | up to 192 hours
  Pharmacokinetic Data Analysis for XZP-3621 and its metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China